CLINICAL TRIAL: NCT05807425
Title: Sclerotherapy With Polidocanol Foam in the Treatment of First, Second and Third-Grade Hemorrhoidal Disease in Patients With Liver Cirrhosis: A Prospective, Cohort Trial
Brief Title: Polidocanol Foam in Hemorrhoidal Disease in Patients With Liver Cirrhosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Paulo Sérgio Durão Salgueiro, Principal investigator, Universidade do Porto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021.051(041-DEFI/042-CE)
Record Dates: First submitted 2023-03-21; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Hemorrhoids; Liver Cirrhosis
Keywords: Hemorrhoids; Liver Cirrhosis; Sclerotehrapy; Polidocanol foam
MeSH Terms: conditions — Hemorrhoids; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: During the intervention period the participants are observed at 3-week intervals (maximum of 3 sessions). The required number of sessions (maximum of 3) is determined by clinical and anoscopic evaluation (if the participant is non-symptomatic and/or there is no significant hemorrhoidal disease on anoscopy, the patient will not be a candidate for additional instrumental therapy moving directly to the follow-up period). After the intervention period, a one-year follow-up is scheduled with medical appointments performed every 3 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polidocanol foam sclerotherapy (Experimental): A cohort of cirrhotic patients with hemorrhoidal disease will be treated with polidocanol foam sclerotherapy.
  Interventions: Procedure: Polidocanol foam sclerotherapy

INTERVENTIONS:
Procedure: Polidocanol foam sclerotherapy — The preparation of the foam is done according to the Tessari's technique using 2 disposable 20ml syringe, a three-way tap and a 10cm reusable extender adapted to intravenous needle. The sclerosant is applied according to the Blanchard's technique through a disposable transparent anoscope with the patient in jack-knife (knee-chest) position. In each session treatment can be performed on more than one hemorrhoidal cushion. The maximum dose per treatment session is 20ml (mixture of 4ml of polidocanol 3% with 16ml of air).

SUMMARY:
Hemorrhoidal disease (HD) is a common health problem, affecting up to 38,9% of adult population. HD is also a common finding in up to 36% of cirrhotic patients, as hemorrhoidal plexus is a possible site of portosystemic venous anastomosis. Cirrhotic patients represent a group often neglected in clinical trials so, little is known about the optimal treatment for HD these patients. The objective of this study is to prospectively evaluate the efficacy and safety of treatment of grade I, II and III internal HD with polidocanol foam in cirrhotic patients.

DETAILED DESCRIPTION:
Hemorrhoidal disease (HD) is a common health problem, affecting up to 38,9% of adult population. Despite being a benign condition, associated symptoms like bleeding, pain, prolapsing, swelling, itching, and mucus soiling impact considerably on patients' quality of life. HD is also a common finding in up to 36% of cirrhotic patients, as hemorrhoidal plexus is a possible site of portosystemic venous anastomosis. Despite portal hypertension does not increase the prevalence of hemorrhoids, elevated portal venous pressure, with a not so rare contribution of coagulopathy, may result in massive, life-threatening hemorrhoidal bleeding, unlike the normal population. Besides, internal HD bleeding is the most frequently identified cause of bleeding with origin on the lower gastrointestinal tract among cirrhotic patients with severe hematochezia .

HD treatment can be grouped into conservative (diet, lifestyle changes, laxatives, anti-inflammatory drugs, phlebotonics), office-based (sclerotherapy, ligation, photocoagulation, laser photocoagulation, among others) and surgical (hemorrhoidectomy, hemorrhoidopexy). The choice of therapy should be oriented by the Goligher's classification, or a symptom score such as Rørvik's Hemorrhoidal Disease Symptom Score (HDSS).

Cirrhotic patients represent a group often neglected in clinical trials so, little is known about the optimal treatment for HD these patients. Surgical treatment with stapled hemorrhoidopexy has been described in cirrhotic patients as a feasible and safe approach, but with up to 46,7% of the procedures complicated with postoperative staple-line bleeding, although all of them managed with conservative treatment without reoperation or death. Recently, Ashraf et al compared hemorrhoidectomy performed using rubber band ligation (RBL) with conventional hemorrhoidectomy in 40 randomized patients with liver disease and diagnosed with grade I, II, or III HD. Intraoperative blood loss was lower in RBL group (1.2 ± 1.6 ml vs 22.2 ± 6.58 ml, p=0,001), as well as operative time (9.00 ± 2.449 min vs 24.100 ± 3.669 min, p=0,001). Importantly, postoperative pain (35% vs 100%, p=0,001), bleeding (15% vs 45%, p=0,022) and urine retention (20% vs 55%, p=0,011) were lower in the RBL group, along with time of hospital stay (8.6 ± 2.54 h vs 60.65 ± 41.93, p=0,002) and time of wound healing (16.85 ± 1.87 days vs 31.00 ± 3.57 days, p=0,003).

Bearing in mind the high rate of surgical complications in cirrhotic patients, these results suggest that office-based treatments, may be the preferred treatment for cirrhotic patients with HD grades I to III. Awad et al, compared the efficacy of endoscopic injection sclerotherapy (EIS) to RBL in the treatment of bleeding internal hemorrhoids in 120 adult patients with liver cirrhosis. Both techniques were highly effective in the control of bleeding with a low rebleeding [10% in the EBL group and 13.33% in the EIS group] and recurrence [20% in the EBL group and 20% in the EIS group] rates; also, EBL had significantly less pain and higher patient satisfaction than EIS. However, these authors have used liquid sclerosing agents (either ethanolamine oleate 5% or N-butyl cyanoacrylate). A recent portuguese study by Fernandes et al has evaluated the efficacy and safety of a sclerosing agent, polidocanol, foam injection in 2000 consecutive patients with prolapsed hemorrhoids (grades II/III/IV). This technique showed high efficacy (98%) and tolerability (92% with mild/no pain) with only 0,7% of serious complications (major bleeding n=3; urinary retention n=4; infection/suppuration requiring surgery n=2). Also, in this cohort, 210 patients (10,5%) were under anticoagulation or double antiplatelet therapy) and only 2 of these patients presented clinically significant bleeding. The authors conclude that polidocanol foam should be used as first-line treatment of most hemorrhoid patient, including those under anticoagulation and antiplatelet therapy. Nevertheless, no cirrhotic patients were included, so results cannot be generalized to this particular high-risk group.

The objective of this study is to prospectively evaluate the efficacy and safety of treatment of grade I, II and III internal hemorrhoidal disease with polidocanol foam in cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with liver cirrhosis and symptomatic HD grades I to III
* Refractory to conservative therapy (dietary modification, intestinal transit modifiers, topical and phlebotonics), during a period of 4 weeks

Exclusion Criteria:

* Known allergy to polidocanol
* Pregnant and lactating women
* Inflammatory bowel disease
* Other concomitant symptomatic perianal disease
* History of office-based or surgical treatment of hemorrhoidal disease in the last 6 months
* Immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Therapeutic success | 9 weeks
  For efficacy evaluation during the intervention period the outcome of therapeutic success (improvement of HDSS) will be assessed; the therapeutic success is subdivided in: complete (HDSS = 0), partial (HDSS > 0 but with improvement over the initial score) or unsuccess (participants that, after 3 sessions of office-based treatment worsened or maintained the initial HDSS
Incidence of Treatment Adverse Events | 9 weeks
  Complications will be assessed and classified as: mild (e.g. pain/discomfort, minor bleeding, external hemorrhoidal thrombosis not requiring surgical intervention); moderate (e.g. external hemorrhoidal thrombosis requiring surgical intervention, moderate bleeding not requiring blood transfusion, urgent hemostasis or urgent surgery); and severe (e.g. sepsis, Fournier's gangrene, perineal abscess, bleeding with hemodynamic instability, transfusion need or urgent surgery, sexual impotence in man).

SECONDARY OUTCOMES:
Variation of Goligher classification (hemorrhoidal prolapse from grade 1 to grade 4) | 9 weeks
  Variation of Goligher classification before and after the intervention
Number of office-based therapy sessions | 9 weeks
  Number of office-based therapy sessions performed during intervention period
Hemorrhoidal disease recurrence | 1 year
  Recurrence during the follow-up period (for patients who have had therapeutic success) will be defined as mild, if HDSS worsened compared to the previous visit but is still better than the initial visit; or severe if HDSS equals or worsens compared to the initial score, requiring instrumental or surgical treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Salgueiro, MD PhD, Principal Investigator — Centro Hospitalar Universitário de Santo António
Locations (1):
- Centro Hospitalar Universitário do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Misra SP, Dwivedi M, Misra V. Prevalence and factors influencing hemorrhoids, anorectal varices, and colopathy in patients with portal hypertension. Endoscopy. 1996 May;28(4):340-5. doi: 10.1055/s-2007-1005477. PMID 8813499
- [Background] Riss S, Weiser FA, Schwameis K, Riss T, Mittlbock M, Steiner G, Stift A. The prevalence of hemorrhoids in adults. Int J Colorectal Dis. 2012 Feb;27(2):215-20. doi: 10.1007/s00384-011-1316-3. Epub 2011 Sep 20. PMID 21932016
- [Background] Hosking SW, Smart HL, Johnson AG, Triger DR. Anorectal varices, haemorrhoids, and portal hypertension. Lancet. 1989 Feb 18;1(8634):349-52. doi: 10.1016/s0140-6736(89)91724-8. PMID 2563507
- [Background] Jacobs DM, Bubrick MP, Onstad GR, Hitchcock CR. The relationship of hemorrhoids to portal hypertension. Dis Colon Rectum. 1980 Nov-Dec;23(8):567-9. doi: 10.1007/BF02988998. PMID 6970115
- [Background] Camus M, Khungar V, Jensen DM, Ohning GV, Kovacs TO, Jutabha R, Ghassemi KA, Machicado GA, Dulai GS. Origin, Clinical Characteristics and 30-Day Outcomes of Severe Hematochezia in Cirrhotics and Non-cirrhotics. Dig Dis Sci. 2016 Sep;61(9):2732-40. doi: 10.1007/s10620-016-4198-y. Epub 2016 Jun 10. PMID 27286877
- [Background] Hull TL. Surgery of the anus, rectum and colon. Gastroenterology. 2000 Oct;119(4):1173-5. doi: 10.1016/s0016-5085(00)80038-4. No abstract available. PMID 11040208
- [Background] Rorvik HD, Styr K, Ilum L, McKinstry GL, Dragesund T, Campos AH, Brandstrup B, Olaison G. Hemorrhoidal Disease Symptom Score and Short Health ScaleHD: New Tools to Evaluate Symptoms and Health-Related Quality of Life in Hemorrhoidal Disease. Dis Colon Rectum. 2019 Mar;62(3):333-342. doi: 10.1097/DCR.0000000000001234. PMID 30451751
- [Background] Huang WS, Lin PY, Chin CC, Yeh CH, Hsieh CC, Chang TS, Wang JY. Stapled hemorrhoidopexy for prolapsed hemorrhoids in patients with liver cirrhosis; a preliminary outcome for 8-case experience. Int J Colorectal Dis. 2007 Sep;22(9):1083-9. doi: 10.1007/s00384-007-0271-5. Epub 2007 Mar 2. PMID 17334772
- [Background] Awad AE, Soliman HH, Saif SA, Darwish AM, Mosaad S, Elfert AA. A prospective randomised comparative study of endoscopic band ligation versus injection sclerotherapy of bleeding internal haemorrhoids in patients with liver cirrhosis. Arab J Gastroenterol. 2012 Jun;13(2):77-81. doi: 10.1016/j.ajg.2012.03.008. Epub 2012 Apr 24. PMID 22980596
- [Background] Fernandes V, Fonseca J. Polidocanol Foam Injected at High Doses with Intravenous Needle: The (Almost) Perfect Treatment of Symptomatic Internal Hemorrhoids. GE Port J Gastroenterol. 2019 May;26(3):169-175. doi: 10.1159/000492202. Epub 2018 Aug 31. PMID 31192285
- [Background] Salgueiro P, Garrido M, Santos RG, Pedroto I, Castro-Pocas FM. Polidocanol Foam Sclerotherapy Versus Rubber Band Ligation in Hemorrhoidal Disease Grades I/II/III: Randomized Trial. Dis Colon Rectum. 2022 Jul 1;65(7):e718-e727. doi: 10.1097/DCR.0000000000002117. Epub 2022 Nov 22. PMID 34840294
- [Background] Salgueiro P, Rei A, Garrido M, Rosa B, Oliveira AM, Pereira-Guedes T, Morais S, Castro-Pocas F. Polidocanol foam sclerotherapy in the treatment of hemorrhoidal disease in patients with bleeding disorders: a multicenter, prospective, cohort study. Tech Coloproctol. 2022 Aug;26(8):615-625. doi: 10.1007/s10151-022-02600-5. Epub 2022 Feb 25. PMID 35217937
- [Background] Neves S, Falcao D, Povo A, Castro-Pocas F, Oliveira J, Salgueiro P. 3% polidocanol foam sclerotherapy versus hemorrhoidal artery ligation with recto anal repair in hemorrhoidal disease grades II-III: a randomized, pilot trial. Rev Esp Enferm Dig. 2023 Mar;115(3):115-120. doi: 10.17235/reed.2022.8568/2022. PMID 35638762
- [Background] Salgueiro P, Ramos MI, Castro-Pocas F, Libanio D. Office-Based Procedures in the Management of Hemorrhoidal Disease: Rubber Band Ligation versus Sclerotherapy - Systematic Review and Meta-Analysis. GE Port J Gastroenterol. 2022 Mar 8;29(6):409-419. doi: 10.1159/000522171. eCollection 2022 Nov. PMID 36545183
- [Background] Salgueiro P, Caetano AC, Oliveira AM, Rosa B, Mascarenhas-Saraiva M, Ministro P, Amaro P, Godinho R, Coelho R, Gaio R, Fernandes S, Fernandes V, Castro-Pocas F. Portuguese Society of Gastroenterology Consensus on the Diagnosis and Management of Hemorrhoidal Disease. GE Port J Gastroenterol. 2020 Feb;27(2):90-102. doi: 10.1159/000502260. Epub 2019 Sep 5. PMID 32266306